CLINICAL TRIAL: NCT03218995
Title: An Open-Label Safety, Tolerability, and Pharmacokinetics Study of Eteplirsen in Young Patients With Duchenne Muscular Dystrophy Amenable to Exon 51 Skipping
Brief Title: Study of Eteplirsen in Young Participants With Duchenne Muscular Dystrophy (DMD) Amenable to Exon 51 Skipping
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4658-102
Record Dates: First submitted 2017-07-09; First posted 2017-07-17 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne; Eteplirsen; dystrophy; dystrophin; exon 51
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eteplirsen (Experimental): Eteplirsen will be administered once every 7 days by intravenous (IV) infusion starting on Day 1 for up to 96 weeks. The starting dose will be 2 milligrams/kilogram (mg/kg) eteplirsen, with escalation to 4, 10, 20, and 30 mg/kg for 10 weeks, and then participants will continue to receive eteplirsen at 30 mg/kg for the duration of the study.
  Interventions: Drug: Eteplirsen

INTERVENTIONS:
Drug: Eteplirsen — Infusion for intravenous use.
  Other Names: AVI-4658; EXONDYS 51®

SUMMARY:
This is a multicenter, open-label, dose-escalation study to evaluate the safety, tolerability, and PK of once-weekly IV infusions of eteplirsen in approximately 12 male participants, ages 6 months to 48 months (inclusive), who have genotypically confirmed DMD with a deletion mutation amenable to exon 51 skipping.

ELIGIBILITY:
Inclusion Criteria:

* Male between 6 months to 48 months of age (inclusive)
* Diagnosis of DMD with a deletion mutation amenable to exon 51 skipping
* Parent(s) or legal guardian(s) who is willing to provide written informed consent

Exclusion Criteria:

* Received treatment that might have an effect on muscle strength or function within 12 weeks prior to dosing
* Received previous or current treatment with any experimental treatment
* Clinically significant illness other than DMD
* Clinically significant laboratory abnormality
* Any other condition that could interfere with the participation in the study.

Ages: 6 Months to 48 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Sarepta Therapeutics, Inc.
Locations (4):
- Universitair ziekenhuis Gent, Ghent, Belgium
- Armand-Trousseau Hospital, Paris, France
- Site Fondazione Policlinico Universitario Agostino Gemelli, Roma, Italy
- UCL Great Ormond Street Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercuri E, Seferian AM, Servais L, Deconinck N, Stevenson H, Ni X, Zhang W, East L, Yonren S, Muntoni F; 4658-102 Study Group. Safety, tolerability and pharmacokinetics of eteplirsen in young boys aged 6-48 months with Duchenne muscular dystrophy amenable to exon 51 skipping. Neuromuscul Disord. 2023 Jun;33(6):476-483. doi: 10.1016/j.nmd.2023.03.008. Epub 2023 Mar 24. PMID 37207382

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with genotypically confirmed Duchenne muscular dystrophy (DMD) featuring a deletion mutation amenable to exon 51 skipping were enrolled into 2 cohorts based on their age.
Groups:
- Eteplirsen: Eteplirsen was administered once every 7 days by intravenous (IV) infusion starting on Day 1 for up to 96 weeks. The starting dose was 2 milligrams/kilogram (mg/kg) eteplirsen, with escalation to 4, 10, 20, and 30 mg/kg for 10 weeks, and then participants continued to receive eteplirsen at 30 mg/kg for the duration of the study.
Period: Overall Study
Arm/Group | Eteplirsen
Started | 15
Received at Least 1 Dose of Study Drug | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study.
Groups:
- Overall Study: Eteplirsen was administered once every 7 days by IV infusion starting on Day 1 for up to 96 weeks. The starting dose was 2 mg/kg eteplirsen, with escalation to 4, 10, 20, and 30 mg/kg for 10 weeks, and then participants continued to receive eteplirsen at 30 mg/kg for the duration of the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: months] | 28.5 (12.94) [lower limit 12.94]
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 6
  Children (2-11 years) | 9
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 0
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity data are reported as "Missing" for participants from France because French sites and the French Regulations prohibit the entry of race and ethnicity.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 7
    Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data are reported as "Missing" for participants from France because French sites and the French Regulations prohibit the entry of race and ethnicity.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 9
    More than one race | 1
    Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and TEAEs Leading to Discontinuation From Study Drug
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. An AE was any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the study drug. Abnormalities presented at Baseline were considered AEs if they reoccurred after resolution or worsen during the AE collection period. An SAE was defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Adverse Events' Section.
Time Frame: Baseline up to Week 100
Population: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Age 24 to 48 Months: Participants aged 24 to 48 months old were administered eteplirsen once every 7 days by IV infusion starting on Day 1 for up to 96 weeks. The starting dose was 2 mg/kg eteplirsen, with escalation to 4, 10, 20, and 30 mg/kg for 10 weeks, and then participants continued to receive eteplirsen at 30 mg/kg for the duration of the study.
- Cohort 2: Age 6 to <24 Months: Participants aged 6 to <24 months old were administered eteplirsen once every 7 days by IV infusion starting on Day 1 for up to 96 weeks. The starting dose was 2 mg/kg eteplirsen, with escalation to 4, 10, 20, and 30 mg/kg for 10 weeks, and then participants continued to receive eteplirsen at 30 mg/kg for the duration of the study.
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
Participants
  TEAE | 9 | 6
  SAE | 0 | 1
  AE leading to discontinuation from study drug | 0 | 0

2. Primary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Clinical Safety Laboratory Abnormality
Description: Clinical laboratory parameters that were evaluated included
  * Any Grade ≥2 (moderate) or serious event without an alternative etiology that the Investigator deemed was related to study drug
  * Two consecutive drug-related serum creatinine levels ≥2*upper limit of normal (ULN) without an alternative etiology
  * Creatine kinase (CK) levels >50,000 units/liter (U/L)
  * A confirmed, unexplained, increase in gamma glutamyl transferase (GGT) >3*ULN and either an increase in bilirubin >2*ULN or nascent prothrombin time >2*ULN concurrently, without an alternative etiology
Time Frame: Baseline up to Week 100
Population: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
Participants | 9 | 6

3. Primary Outcome: Number of Participants With at Least 1 Markedly Abnormal Vital Sign
Description: The vital sign parameters that were evaluated included blood pressure, heart rate, respiration, and temperature. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Adverse Events' Section.
Time Frame: Baseline up to Week 100
Population: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
Participants | 9 | 6

4. Primary Outcome: Abnormal Changes From Baseline or Worsening of Physical Examination Findings
Description: Data not collected during the study for this Outcome Measure. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Adverse Events' Section.
Time Frame: Baseline up to Week 100
Population: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study. Data were not collected for this Outcome Measure.
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Number of Participants With at Least 1 Markedly Abnormal Electrocardiogram (ECG) and Echocardiogram (ECHO)
Description: The ECG was manually reviewed and interpreted by medically qualified personnel using a central vendor according to pre-specified criteria. The Investigator determined if the findings in the centrally read ECG report were clinically significant. Clinical significance was defined as any variation in ECG findings that had medical relevance resulting in an alteration in medical care. The ECHO was reviewed and interpreted by medically qualified personnel using a central vendor according to pre-specified criteria. The Investigator determined if the findings in the ECHO report were clinically significant. Clinical significance was defined as any variation in ECHO findings that had medical relevance resulting in an alteration in medical care. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in the 'Adverse Events' Section.
Time Frame: Weeks 8, 12, 24, 36, 48, 60, 72, 84, 96
Population: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
Participants | 4 | 5

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Eteplirsen
Time Frame: Pre-infusion, immediately prior to end of infusion, and approximately 1-3 hours and 6-8 hours after completion of infusion during Weeks 2 (2 mg/kg dose level), 6 (10 mg/kg dose level), 8 (20 mg/kg dose level), and 10 and 24 (30 mg/kg dose level)
Population: The Safety Set was used for pharmacokinetic(s) (PK) analysis and included all participants who were enrolled and received at least 1 dose of eteplirsen during the study. PK data were not collected for participants who received 4 mg of eteplirsen. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
microgram/milliliter (μg/mL)
  Week 2 (2 mg/kg): number analyzed (Participants) | 8 | 5
  Week 2 (2 mg/kg) | 9.67 (75.9) | 4.22 (120)
  Week 6 (10 mg/kg) | 46.5 (72.3) | 17.2 (192)
  Week 8 (20 mg/kg) | 63.3 (123) | 85.0 (67.6)
  Week 10 (30 mg/kg) | 93.7 (55.5) | 63.8 (124)
  Week 24 (30 mg/kg): number analyzed (Participants) | 8 | 6
  Week 24 (30 mg/kg) | 78.2 (92.2) | 59.7 (82.7)

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Eteplirsen
Time Frame: as for outcome 6
Population: The Safety Set was used for PK analysis and included all participants who were enrolled and received at least 1 dose of eteplirsen during the study. PK data were not collected for participants who received 4 mg of eteplirsen. Here, 'Number Analyzed' signifies number of participants evaluable at the specified timepoint.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
hours (hr)
  2 mg/kg (Week 2): number analyzed (Participants) | 8 | 5
  2 mg/kg (Week 2) | 0.58 [0.17 to 2.67] | 0.58 [0.42 to 0.67]
  10 mg/kg (Week 6) | 0.58 [0.47 to 4.25] | 0.72 [0.58 to 3.32]
  20 mg/kg (Week 8) | 0.78 [0.50 to 2.75] | 0.73 [0.53 to 1.17]
  30 mg/kg (Week 10) | 0.58 [0.50 to 1.48] | 0.92 [0.50 to 2.75]
  30 mg/kg (Week 24): number analyzed (Participants) | 8 | 6
  30 mg/kg (Week 24) | 0.63 [0.42 to 6.83] | 0.72 [0.58 to 1.83]

8. Secondary Outcome: Area Under Concentration-Time Curve From Time 0 to the Last Quantifiable Concentration (AUClast) of Eteplirsen in Plasma
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
μg*hr/mL
  2 mg/kg (Week 2): number analyzed (Participants) | 8 | 5
  2 mg/kg (Week 2) | 13.8 (118) | 6.13 (73.1)
  10 mg/kg (Week 6) | 56.1 (57.2) | 27.8 (113)
  20 mg/kg (Week 8) | 92.1 (94.7) | 81.4 (89.6)
  30 mg/kg (Week 10) | 119 (30.8) | 85.0 (114)
  30 mg/kg (Week 24): number analyzed (Participants) | 8 | 6
  30 mg/kg (Week 24) | 100 (42.5) | 89.6 (43.8)

9. Secondary Outcome: Amount of Drug Eliminated in Urine
Description: Amount of unchanged drug excreted in urine from time 0 to 4 hours after completion of dosing is reported.
Time Frame: as for outcome 6
Population: The Safety Set was used for PK analysis and included all participants who were enrolled and received at least 1 dose of eteplirsen during the study. PK data were not collected for participants who received 4 mg of eteplirsen. Here, 'Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
Number analyzed (Participants) | 9 | 6
μg
  2 mg/kg dose (Week 2): number analyzed (Participants) | 3 | 3
  2 mg/kg dose (Week 2) | 7720 (9060) | 1430 (1390)
  10 mg/kg (Week 6): number analyzed (Participants) | 7 | 6
  10 mg/kg (Week 6) | 56000 (73300) | 28700 (24100)
  20 mg/kg (Week 8): number analyzed (Participants) | 6 | 5
  20 mg/kg (Week 8) | 102000 (108000) | 65600 (47900)
  30 mg/kg (Week 10): number analyzed (Participants) | 8 | 6
  30 mg/kg (Week 10) | 263000 (209000) | 94700 (68500)
  30 mg/kg (Week 24): number analyzed (Participants) | 7 | 4
  30 mg/kg (Week 24) | 239000 (140000) | 147000 (132000)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 100
Description: The Safety Set included all participants who were enrolled and received at least 1 dose of eteplirsen during the study.
Arm/Group | Cohort 1: Age 24 to 48 Months | Cohort 2: Age 6 to <24 Months
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Age 24 to 48 Months (N=9) | Cohort 2: Age 6 to <24 Months (N=6)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Age 24 to 48 Months (N=9) | Cohort 2: Age 6 to <24 Months (N=6)
Nasopharyngitis (Infections and infestations) | 7 (27) | 5 (19)
Rhinitis (Infections and infestations) | 4 (4) | 4 (9)
Ear infection (Infections and infestations) | 3 (6) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (6) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4)
Eye infection (Infections and infestations) | 0 (0) | 1 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (2)
Roseola (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (21) | 6 (21)
Catheter site eczema (General disorders) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 8 (15) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 3 (9)
Constipation (Gastrointestinal disorders) | 2 (8) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 2 (5)
Head injury (Injury, poisoning and procedural complications) | 5 (7) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (25) | 5 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (9) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (8)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inner ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyposideraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 1 (3) | 1 (2)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Body temperature (Investigations) | 1 (3) | 1 (1)
Body temperature increased (Investigations) | 1 (2) | 1 (3)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0)
Haemophilus test positive (Investigations) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Autoimmune neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemoglobinopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Allergy to chemicals (Immune system disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03218995/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03218995/SAP_001.pdf